CLINICAL TRIAL: NCT05301088
Title: The Effect of Chocolate Smell and Stress Ball on Pain and Fear in Venous Blood Collection in Children
Brief Title: Pain and Fear of Venous Blood Collection in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Eylem Nazan KAPAN (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, PhD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.O.O.0l 0/184
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Pain; Fear
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chocolate Scent (Experimental)
  Interventions: Other: Chocolate Scent
- Stress Ball (Experimental)
  Interventions: Other: Chocolate Scent
- Control (No Intervention)

INTERVENTIONS:
Other: Chocolate Scent — Chocolate Scent:Children in this group will be given chocolate scent sniffing as a non-pharmacological distraction method.
  Stress Ball:Stress ball squeezing will be used as a non-pharmacological distraction method for children in this group.
  Other Names: Stress Ball
  Arms: Chocolate Scent; Stress Ball

SUMMARY:
Nurses are in the position of primary health care provider in relieving children's pain and fears of bloodletting in the wards where they work. As a result of this study, it is aimed to encourage nurses to apply non-pharmacological interventions during painful medical procedures, to facilitate the provision of necessary and different means of distraction to blood collection services, and to contribute to the development of in-house health policies and the preparation of appropriate clinical guides and to add an innovative perspective.

ELIGIBILITY:
Inclusion Criteria:

* 6-12 age group,
* children who need blood drawn for any reason
* have no disease that can cause chronic pain,
* no olfactory disorder
* no mental or neurological problems
* able to communicate
* speaks Turkish

Exclusion Criteria:

* those who did not give consent to the research by both the child and the parent

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Rating Scale | 12 week
Child Fear Scale | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)